CLINICAL TRIAL: NCT06468878
Title: The Influence of Music on Response to Virtual Reality-Based Exposure for Acrophobia
Brief Title: Virtual Reality Intervention for Fear of Heights
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7169E
Record Dates: First submitted 2024-06-16; First posted 2024-06-21 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Acrophobia
MeSH Terms: conditions — Acrophobia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure Intervention with Non-Lyrical, Liked Background Music (Experimental): Participants will be presented with a list of instrumental songs without lyrics from popular movies. Participants will then rank the songs in order of those they would like to hear the most. During VR heights exposure the participants' highest-ranked songs will be played in the background at a low volume.
  Interventions: Behavioral: Exposure Intervention Plus Music Induction
- Exposure Intervention without Background Music (Experimental): Participants will undergo VR heights exposure without background music.
  Interventions: Behavioral: Exposure Intervention With No Music Induction

INTERVENTIONS:
Behavioral: Exposure Intervention Plus Music Induction — VR exposure for acrophobia with background music.
  Arms: Exposure Intervention with Non-Lyrical, Liked Background Music
Behavioral: Exposure Intervention With No Music Induction — VR exposure for acrophobia with no background music.
  Arms: Exposure Intervention without Background Music

SUMMARY:
Exposure-based cognitive behavior therapy is an efficacious treatment for acrophobia (fear of heights) and has been delivered effectively in a virtual reality (VR) environment. The present study is designed to evaluate the effects of liked, non-lyrical background music on the efficacy of a brief VR exposure intervention.

DETAILED DESCRIPTION:
The goal of this clinical trial is to compare acrophobia (fear of heights) outcomes for VR exposure therapy in college students with elevated acrophobia when listening to music during exposure versus no music. The overarching aim of the current study is to determine how liked, non-lyrical background music will influence acrophobia outcomes after a brief exposure therapy session in VR.

The study involves three phases: (1) initial screening, (2) in-person assessment and a brief exposure intervention for a subset of participants with elevated acrophobia, and (3) a one-week follow-up assessment conducted online. Students who choose to participate and screen high on an acrophobia scale will be assigned to an experimental or control condition prior to undergoing VR based exposure therapy. Acrophobia outcomes are measured immediately post-intervention and one week later.

Researchers will compare participants in the music condition to participants in the non-music condition to see if acrophobia outcomes differ.

ELIGIBILITY:
Inclusion Criteria:

* Self-report of 18 years of age or older
* Current student at Boston University
* Ability to read English to provide informed consent
* Familiarity with a computer keyboard and mouse or a touch screen device (e.g. phone, tablet)
* For Phase 2: Acrophobia score of ≥ 45.45 on the Acrophobia Questionnaire (AQ) Anxiety Subscale

Exclusion Criteria:

* Previous participation (i.e. no participant may take the survey more than once).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Acrophobia (Fear of Heights) | Comparison of pre-exposure scores to scores from the follow-up survey one week after exposure
  Assessed using the Acrophobia Questionnaire (AQ) Anxiety Subscale

SECONDARY OUTCOMES:
Valance | Comparison of pre-exposure scores to scores from the follow-up survey one week after exposure
  Self-report measure of how participant feels about experiencing high-height environments.
Height-Relevant Interpretations | Comparison of pre-exposure scores to scores from the follow-up survey one week after exposure
  Assessed using the Heights Interpretation Questionnaire (HIQ)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Long, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No